CLINICAL TRIAL: NCT00130897
Title: A SU011248 Expanded Access Protocol For Systemic Therapy Of Patients With Metastatic Renal Cell Carcinoma Who Are Ineligible For Participation In Other SU011248 Protocols But May Derive Benefit From Treatment With SU011248
Brief Title: Treatment Use Study With Sunitinib (SU011248) For Patients With Cytokine-Refractory Metastatic Renal Cell Carcinoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181037
Record Dates: First submitted 2005-08-14; First posted 2005-08-16 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

INTERVENTIONS:
Drug: Sutent — Sutent, 25, 37.5. or 50 mg daily

SUMMARY:
The primary objective of this protocol is to provide access to SU011248 treatment for patients with metastatic RCC who are ineligible for participation in ongoing SU011248 clinical studies and have the potential to derive clinical benefit from treatment with SU011248 based on the judgment of the investigator.

DETAILED DESCRIPTION:
Given that an Expanded Access study does not meet the definition of a controlled clinical investigation, and as such, is not considered an applicable drug clinical trial per NIH, Basic Results for such studies are not required to be reported. Protocol A6181037 has been identified as an Expanded Access trial, and has been registered to ClinicalTrials.gov, however Basic Results will not be posted.

ELIGIBILITY:
Inclusion Criteria:

* renal cell carcinoma that is not amendable to standard therapy with curative intent

Exclusion Criteria:

* current treatment in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (228):
- United States (38):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Council Bluffs, Iowa
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Pfizer Investigational Site, Buenos Aires, Argentina
- Australia (9):
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, South Brisbane, Queensland
  - Pfizer Investigational Site, Elizabeth Vale, South Australia
  - Pfizer Investigational Site, Woodville South, South Australia
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, Heidelburg, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
- Belgium (5):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Wilrijk
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- Brazil (6):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Jaú, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (2):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Sofia
- Canada (13):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Winnnipeg, Manitoba
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Santiago, RM, Chile
- Colombia (2):
  - Pfizer Investigational Site, Bogotá, Cundinamarca
  - Pfizer Investigational Site, Cali
- Croatia (2):
  - Pfizer Investigational Site, Rijeka
  - Pfizer Investigational Site, Split
- Czechia (3):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Prague
- Ecuador (2):
  - Pfizer Investigational Site, Guayaquil, Guayas
  - Pfizer Investigational Site, Quito, Pichincha
- Egypt (2):
  - Pfizer Investigational Site, Cairo
  - Pfizer Investigational Site, Giza
- Pfizer Investigational Site, Turku, Finland
- France (12):
  - Pfizer Investigational Site, Lyon, Cedex 08
  - Pfizer Investigational Site, Saint-Herblain, Cedex
  - Pfizer Investigational Site, Strasbourg, Cedex
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Clermont Ferand
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Rostock
  - Pfizer Investigational Site, Ulm
- Greece (4):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
- Pfizer Investigational Site, Hong Hong, Hong Kong, Hong Kong
- Pfizer Investigational Site, Budapest, Hungary
- India (5):
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Pārel, Mumbai
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, New Delhi
- Pfizer Investigational Site, Dublin, Ireland
- Israel (2):
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (15):
  - Pfizer Investigational Site, Bergamo
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Cattolica (RN)
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Legnago, VR
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pordenone
  - Pfizer Investigational Site, Rimini
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
- Pfizer Investigational Site, Beirut, Lebanon
- Malaysia (2):
  - Pfizer Investigational Site, Petaling Jaya, Selangor
  - Pfizer Investigational Site, Kuala Lumpur
- Mexico (6):
  - Pfizer Investigational Site, Chihuahua City, Chihuahua
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Puebla City, Puebla
  - Pfizer Investigational Site, Toluca, State of Mexico
  - Pfizer Investigational Site, Mérida, Yucatán
- Netherlands (4):
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Groningen, Provincie Groningen
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Rotterdam
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Panama City, Provincia de Panamá, Panama
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Pfizer Investigational Site, Quezon City, Philippines
- Poland (5):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (2):
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Romania (2):
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Cluj-Napoca
- Russia (3):
  - Pfizer Investigational Site, Obninsk, Kaluga Oblast
  - Pfizer Investigational Site, Chelyabinsk
  - Pfizer Investigational Site, Moscow
- Pfizer Investigational Site, Belgrade, Serbia
- Pfizer Investigational Site, Singapore, Singapore
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Žilina
- Pfizer Investigational Site, Ljubljana, Ljubljana, Slovenia
- Pfizer Investigational Site, Seoul, South Korea
- Spain (10):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'hospitalet Del Llobregat, Barcelona
  - Pfizer Investigational Site, A Coruña, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Salamanca, Salamanca
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Barakaldo, Vizcaya
- Sweden (4):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Umeå
- Switzerland (9):
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bellinzona
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Biel
  - Pfizer Investigational Site, Ch-4058 Basel
  - Pfizer Investigational Site, Ch-4101 Bruderholz
  - Pfizer Investigational Site, Ch-4410 Liesthal
  - Pfizer Investigational Site, Chur
  - Pfizer Investigational Site, Geneva
- Taiwan (2):
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taoyun
- Pfizer Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Istanbul, Capa
  - Pfizer Investigational Site, Istanbul, Cerrahpasa
- United Kingdom (17):
  - Pfizer Investigational Site, Whitchurch, Cardiff
  - Pfizer Investigational Site, London, Se1 9rt
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Leeds, West Yorkshire
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Cottingham
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Guildford
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Northwood
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Swansea
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, Distrito Federal
  - Pfizer Investigational Site, Caracas, Miranda

REFERENCES:
- [Derived] Barrios CH, Herchenhorn D, Chacon M, Cabrera-Galeana P, Sajben P, Zhang K. Safety and efficacy of sunitinib in patients from Latin America: subanalysis of an expanded access trial in metastatic renal cell carcinoma. Onco Targets Ther. 2016 Sep 23;9:5839-5845. doi: 10.2147/OTT.S109445. eCollection 2016. PMID 27713637
- [Derived] Lee SH, Bang YJ, Mainwaring P, Ng C, Chang JW, Kwong P, Li RK, Sriuranpong V, Toh CK, Yuan J, Pitman Lowenthal S, Chung HC. Sunitinib in metastatic renal cell carcinoma: an ethnic Asian subpopulation analysis for safety and efficacy. Asia Pac J Clin Oncol. 2014 Sep;10(3):237-45. doi: 10.1111/ajco.12163. Epub 2014 Feb 27. PMID 24576311
- [Derived] Gore ME, Hariharan S, Porta C, Bracarda S, Hawkins R, Bjarnason GA, Oudard S, Lee SH, Carteni G, Nieto A, Yuan J, Szczylik C. Sunitinib in metastatic renal cell carcinoma patients with brain metastases. Cancer. 2011 Feb 1;117(3):501-9. doi: 10.1002/cncr.25452. Epub 2010 Sep 22. PMID 20862748
- [Derived] Gore ME, Szczylik C, Porta C, Bracarda S, Bjarnason GA, Oudard S, Hariharan S, Lee SH, Haanen J, Castellano D, Vrdoljak E, Schoffski P, Mainwaring P, Nieto A, Yuan J, Bukowski R. Safety and efficacy of sunitinib for metastatic renal-cell carcinoma: an expanded-access trial. Lancet Oncol. 2009 Aug;10(8):757-63. doi: 10.1016/S1470-2045(09)70162-7. Epub 2009 Jul 15. PMID 19615940
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181037&StudyName=Treatment%20Use%20Study%20With%20Sunitinib%20%28SU011248%29%20For%20Patients%20With%20Cytokine-Refractory%20Metastatic%20Renal%20Cell%20Carcinoma